CLINICAL TRIAL: NCT03335085
Title: Long-term Consequences of Childhood Adversity: Exploring Stress Responsive Molecular Pathways and Psychobiological Intervention Models
Brief Title: Oxytocin Administration and Emotion Recognition Abilities in Adults Reporting Adverse Childhood Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Prof. Robert Kumsta, Professor of Genetic Psychology, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KU 2479/3-1
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Single dose of intranasally administered 24 IU of Oxytocin (Syntocinon-Spray Novartis, Switzerland)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): All ingredients except for oxytocin.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin
Other: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates whether intranasal administration of a single dose of oxytocin improves the ability to recognize emotional states. In a cross-over design, half of the participants first received oxytocin, the other half first received placebo.

DETAILED DESCRIPTION:
Adverse childhood experience such as neglect or abuse can lead to long-term deficits in emotion processing abilities, and these effects might be mediated via alterations in oxytocin production or sensitivity. The goal of this study was to test whether emotion recognition abilities and empathy might be improved by intranasal oxytocin administration in adults with a history of childhood maltreatment.

In a double-blind, placebo-controlled experiment with a crossover design, we assessed the performance of 40 healthy participants with a history of childhood adversity on the Reading the Mind in the Eyes Test (RMET) and an emotion recognition task under 24 IU oxytocin vs. placebo and compared them to a control group of 40 matched individuals without traumatic childhood experiences.

ELIGIBILITY:
Inclusion Criteria:

• presence of moderate to severe experiences of childhood adversity (early adversity group)

Exclusion Criteria:

* Acute psychiatric disorders and personality disorders or psychiatric disorders within the last 12 months
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2013-03-23 (Actual); Study Completion 2013-11-05 (Actual)

PRIMARY OUTCOMES:
Reading the Mind in the Eyes Test | 45 minutes post-dose
  Requires participants to infer complex mental states fromthe eye region
Gradual Emotion Recognition Test | 50 minutes post-dose
  Requires participants to swiftly and accurately detect basic emotions form naturalistic, animated stimuli.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwaiger M, Heinrichs M, Kumsta R. Oxytocin administration and emotion recognition abilities in adults with a history of childhood adversity. Psychoneuroendocrinology. 2019 Jan;99:66-71. doi: 10.1016/j.psyneuen.2018.08.025. Epub 2018 Aug 27. PMID 30189345